CLINICAL TRIAL: NCT02865850
Title: Phase 3, Randomized, Open-Label, Active-Controlled Study Evaluating the Efficacy and Safety of Oral Vadadustat for the Correction or Maintenance Treatment of Anemia in Subjects With Incident Dialysis-Dependent Chronic Kidney Disease (DD-CKD) (INNO2VATE - CORRECTION/CONVERSION)
Brief Title: Efficacy and Safety Study to Evaluate Vadadustat for the Correction or Maintenance Treatment of Anemia in Participants With Incident Dialysis-dependent Chronic Kidney Disease (DD-CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0016; 2016-000838-21 (EudraCT Number)
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Anemia; Dialysis-Dependent Chronic Kidney Disease
Keywords: Vadadustat; AKB-6548; anemia; chronic kidney disease; CKD; chronic renal insufficiency; renal impairment; erythropoietin; kidney; renal; oral anemia treatment; hemoglobin; hypoxia-inducible factor; HIF; efficacy; safety; phase 3; cardiovascular
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat; Darbepoetin alfa

STUDY DESIGN:
Masking Description: Sponsor was blinded during the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Vadadustat (Experimental)
  Interventions: Drug: Vadadustat
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Vadadustat — Oral dose administered once daily for ≥36 weeks. Dose adjustment based on hemoglobin level as defined in the protocol.
  Other Names: AKB-6548
  Arms: Vadadustat
Drug: Darbepoetin alfa — Subcutaneous or intravenous dose administered for ≥36 weeks. Initial dose based on the current package insert for investigational sites in the United States (US), and the Summary of Product Characteristics for all other investigational sites (non-US) for adult participants with chronic kidney disease not on dialysis. For participants already on Darbepoetin alfa, the initial dosing regimen in the study was based on the prior dosing regimen.
  Other Names: Aranesp
  Arms: Darbepoetin alfa

SUMMARY:
A multicenter, randomized, open-label, active-controlled Phase 3 study for the correction or maintenance treatment of anemia in participants with incident dialysis-dependent chronic kidney disease (DD-CKD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active-controlled Phase 3 study of the efficacy and safety of Vadadustat versus Darbepoetin alfa for the correction or maintenance treatment in participants with anemia secondary to chronic kidney disease who have recently initiated dialysis treatment for end-stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Initiated chronic maintenance dialysis (either peritoneal or hemodialysis) for end-stage kidney disease within 16 weeks prior to Screening
* Mean Screening hemoglobin between 8.0 and <11.0 grams per deciliter (g/dL) (inclusive)
* Serum ferritin ≥100 nanograms per deciliter (ng/mL) and TSAT ≥20% during Screening

Exclusion Criteria:

* Anemia due to a cause other than chronic kidney disease or participants with active bleeding or recent blood loss
* Red blood cells transfusion within 8 weeks prior to randomization
* Anticipated to recover adequate kidney function to no longer require dialysis
* Uncontrolled hypertension
* Severe heart failure at Screening (New York Heart Association Class IV)
* Acute coronary syndrome (hospitalization for unstable angina, myocardial infarction); surgical or percutaneous intervention for coronary, cerebrovascular, or peripheral artery disease (aortic or lower extremity); surgical or percutaneous valvular replacement or repair; sustained ventricular tachycardia; hospitalization for congestive heart failure; or stroke within 12 weeks prior to or during Screening.
* Participants meeting the criteria of erythropoiesis-stimulating agent resistance within 8 weeks prior to or during Screening defined as follows

  1. epoetin: > 7700 units/dose three times per week or >23,000 units per week
  2. Darbepoetin alfa: >100 micrograms per week (mcg/week)
  3. methoxy polyethylene glycol-epoetin beta: >100 micrograms (mcg) every other week or >200 mcg/month
* Hypersensitivity to Vadadustat, Darbepoetin alfa or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (108):
- United States (50):
  - Research Site, Huntsville, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Anaheim, California
  - Research Site, Canyon Country, California
  - Research Site, Downey, California
  - Research Site, Glendale, California
  - Research Site, Granada Hills, California
  - Research Site, La Mesa, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Montebello, California
  - Research Site, Monterey Park, California
  - Research Site, Newhall, California
  - Research Site #1, Northridge, California
  - Research Site #2, Northridge, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Dimas, California
  - Research Site, Whittier, California
  - Research Site, Arvada, Colorado
  - Research Site, Westminster, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Coral Gables, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site #2, Lawrenceville, Georgia
  - Research Site, Statesboro, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Takoma Park, Maryland
  - Research Site, Roseville, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Astoria, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site #1, Chattanooga, Tennessee
  - Research Site #2, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Hampton, Virginia
- Argentina (9):
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Research Site, Junín, Buenos Aires
  - Research Site, Pergamino, Buenos Aires
  - Research Site, Temperley, Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Salta
  - Research Site, San Luis
- Brazil (12):
  - Research Site, Fortaleza, Ceará
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Juiz de Fora, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site, Maringá, Paraná
  - Research Site, Canoas, Rio Grande do Sul
  - Research Site, Passo Fundo, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Joinville, Santa Catarina
  - Research Site, Santo André, São Paulo
  - Research Site, São Bernardo do Campo, São Paulo
  - Research Site, São Paulo, São Paulo
- Germany (3):
  - Research Site, Villingen-Schwenningen, Baden-Wurttemberg
  - Research Site, Rostock, Mecklenburg-Vorpommern
  - Research Site, Düsseldorf, North Rhine-Westphalia
- Italy (7):
  - Research Site, San Giovanni Rotondo, Foggia
  - Research Site, Genova
  - Research Site, Lecco
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Siena
- Mexico (3):
  - Research Site, Zapopan, Jalisco
  - Research Site, Morelia, Michoacán
  - Research Site, Culiacán, Sinaloa
- Poland (2):
  - Research Site, Golub-Dobrzyń
  - Research Site, Lodz
- Portugal (2):
  - Research Site, Leiria
  - Research Site, Loures
- Russia (4):
  - Research Site #2, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Korea (4):
  - Research Site, Chuncheon, Gangwon-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Seoul
- Ukraine (12):
  - Research Site, Brovary
  - Research Site, Cherkassy
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Mykolaiv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chertow GM, Eckardt KU, Sarnak MJ, Winkelmayer WC, Agarwal R, Minga T, Luo W, Burke SK. Safety and Efficacy of Vadadustat for the Treatment of CKD-Related Anemia within and outside the United States. J Am Soc Nephrol. 2025 Oct 1;36(10):1984-1997. doi: 10.1681/ASN.0000000708. Epub 2025 May 13. PMID 40359056
- [Derived] Sarnak MJ, Agarwal R, Boudville N, Chowdhury PCP, Eckardt KU, Gonzalez CR, Kooienga LA, Koury MJ, Ntoso KA, Luo W, Parfrey PS, Vargo DL, Winkelmayer WC, Zhang Z, Chertow GM. Vadadustat for treatment of anemia in patients with dialysis-dependent chronic kidney disease receiving peritoneal dialysis. Nephrol Dial Transplant. 2023 Sep 29;38(10):2358-2367. doi: 10.1093/ndt/gfad074. PMID 37096396
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Eckardt KU, Agarwal R, Aswad A, Awad A, Block GA, Bacci MR, Farag YMK, Fishbane S, Hubert H, Jardine A, Khawaja Z, Koury MJ, Maroni BJ, Matsushita K, McCullough PA, Lewis EF, Luo W, Parfrey PS, Pergola P, Sarnak MJ, Spinowitz B, Tumlin J, Vargo DL, Walters KA, Winkelmayer WC, Wittes J, Zwiech R, Chertow GM. Safety and Efficacy of Vadadustat for Anemia in Patients Undergoing Dialysis. N Engl J Med. 2021 Apr 29;384(17):1601-1612. doi: 10.1056/NEJMoa2025956. PMID 33913638

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 652 participants were screened for entry into the study. Of these, 369 participants were enrolled and randomized in the study.
Groups:
- Vadadustat: Participants were randomized to receive Vadadustat at an initial oral dose of 300 milligrams per day (mg/day). Thereafter, Vadadustat was taken once daily on an outpatient basis. Up-and-down titration to 150, 300, 450, and 600 mg (available tablet strength was administered as the appropriate number of 150 mg tablets) was allowed during the study based on hemoglobin (Hb) level measurements to maintain target Hb levels.
- Darbepoetin Alfa: Participants were randomized to Darbepoetin alfa at an initial dose that was based on the current package insert for investigational sites in the United States (US), and the Summary of Product Characteristics (SmPC) for all other investigational sites (non-US) for adult participants with chronic kidney disease on dialysis. For participants already on Darbepoetin alfa, the initial dosing regimen in the study was based on the prior dosing regimen.
Period: Overall Study
Arm/Group | Vadadustat | Darbepoetin Alfa
Started | 181 | 188
Completed | 160 | 165
Not Completed | 21 | 23
Not completed — Death | 15 | 19
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 181 | 188 | 369
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (14.80) | 55.6 (14.60) | 56.0 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 75 | 149
  Male | 107 | 113 | 220
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 8 | 20
  Black or African American | 38 | 35 | 73
  White | 129 | 143 | 272
  Not Reported | 0 | 1 | 1
  Reported as Other | 0 | 1 | 1
  Multiple | 1 | 0 | 1
Average hemoglobin [Mean (Standard Deviation); unit: Grams per deciliter (g/dL)] | 9.369 (1.0701) | 9.190 (1.1381) | 9.278 (1.1074)
Number of Participants on Different Types of Dialysis [Count of Participants; unit: Participants] — Dialysis assessment was performed at least 12 weeks prior to the first screening visit. A participant could be included for both peritoneal dialysis and hemodialysis at Baseline (i.e., not mutually exclusive parameters). Population: Dialysis assessment was summarized in the Safety Population (INNO2VATE) which included all participants from the INNO2VATE population who received 1 or more doses of study drug.
  Participants
    Peritoneal Dialysis: number analyzed (Participants) | 179 | 186 | 365
    Peritoneal Dialysis | 22 | 16 | 38
    Hemodialysis: number analyzed (Participants) | 179 | 186 | 365
    Hemodialysis | 158 | 169 | 327
    Chronic Dialysis Not Previously Initiated: number analyzed (Participants) | 179 | 186 | 365
    Chronic Dialysis Not Previously Initiated | 1 | 1 | 2
Mean Years Since Chronic Dialysis Initiated [Mean (Standard Deviation); unit: Years] — Population: Participants with missing chronic dialysis initiation date were not included for the analysis.
  Years
    number analyzed (Participants) | 179 | 186 | 365
    (all) | 0.138 (0.0883) | 0.151 (0.2848) | 0.145 (0.2123)
Number of Participants with History of Diabetes [Count of Participants; unit: Participants] | 81 | 82 | 163
Number of Participants with NYHA Functional Classification of Heart Failure [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) functional classification serves as a fundamental descriptor of heart failure. NYHA heart failure classes are as follows: Class 0 (no congestive heart failure [CHF]), Class I (No symptoms and no limitation in ordinary physical activity), Class II (Mild symptoms and slight limitation during ordinary activity), Class III (Marked limitation in activity due to symptoms, even during less-than-ordinary activity), and Class IV (Severe limitations. Experiences symptoms even while at rest). NYHA class IV is also an exclusion criteria.
  Participants
    NYHA Class 0 | 129 | 126 | 255
    NYHA Class I | 30 | 35 | 65
    NYHA Class II | 18 | 23 | 41
    NYHA Class III | 3 | 4 | 7
    NYHA Class IV | 0 | 0 | 0
    NYHA Class Missing | 1 | 0 | 1
Number of Participants with Any History of Heart Failure [Count of Participants; unit: Participants]
  Yes | 16 | 15 | 31
  No | 54 | 62 | 116
  Missing | 111 | 111 | 222

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hb) to the Average Over the Primary Efficacy Period (Weeks 24 to 36)
Description: The Baseline average was calculated as the average of the Hb values obtained at the screening visit closest to the date of randomization and the randomization visit. The average for the Primary Efficacy Period was calculated as the average Hb value over Weeks 24 to 36. Analysis was conducted using an analysis of covariance (ANCOVA) model with multiple imputation for missing data with Baseline hemoglobin concentration (<9.5 versus ≥9.5 g/dL), geographic region (United States [US] versus European Union [EU] versus Rest of World [ROW]), and New York Heart Association congestive heart failure (NYHA CHF) class (Class 0 [no CHF] or I versus II or III) as covariates.
Time Frame: Baseline; Weeks 24 to 36
Population: Randomized Population: All participants randomized. Analyses of this population were based on the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 181 | 188
Grams per deciliter (g/dL) | 1.26 (0.109) | 1.58 (0.108)
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Treatment comparison: Vadadustat minus Darbepoetin Alfa; Test type: Non-Inferiority — Establishment of non-inferiority was based on a margin of -0.75 g/dL applied to the difference in mean change: Vadadustat minus Darbepoetin alfa; Least squares mean difference = -0.31, 95% CI 2-sided [-0.53 to -0.10], Standard Error of Mean 0.11

2. Primary Outcome: Median Time to First Major Adverse Cardiovascular Event (MACE)
Description: MACE was defined as all-cause mortality, non-fatal myocardial infarction (MI), or non-fatal stroke. The primary safety outcome was positively adjudicated first MACE, which was defined as any death, Endpoint Adjudication Committee (EAC)-confirmed non-fatal MI, or EAC-confirmed non-fatal stroke occurring between the first dose date and each participant's last participation date. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0016 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 176 weeks
Population: Safety Population (INNO2VATE): All participants from the INNO2VATE population who received 1 or more doses of study drug. Only those participants with MACE events were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 22 | 24
Weeks | 26.21 [13.71 to 50.00] | 46.64 [22.86 to 58.14]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0016 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per Food and Drug Administration [FDA]) and 1.30 (per European Medicines Agency [EMA]); p = 0.9950, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.536 to 1.761]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first MACE for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 355 and 377 respectively; median time to first event (Q1, Q3) = 46.14 (24.71, 77.14) weeks versus 47.00 (22.43, 74.43) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.4877, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.833 to 1.113]

3. Secondary Outcome: Change From Baseline in Hb to the Average Over the Secondary Efficacy Period (Weeks 40 to 52)
Description: The Baseline average was calculated as the average of the Hb values obtained at the screening visit closest to the date of randomization and the randomization visit. The average for the Secondary Efficacy Period was calculated as the average Hb value over Weeks 40 to 52. Analysis was conducted using an ANCOVA model with multiple imputation for missing data with Baseline hemoglobin concentration (<9.5 versus ≥9.5 g/dL), geographic region (US versus EU versus ROW), and NYHA CHF class (Class 0 [no CHF] or I versus II or III) as covariates.
Time Frame: Baseline; Weeks 40 to 52
Population: Randomized Population. Analyses of this population were based on the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 181 | 188
g/dL | 1.42 (0.132) | 1.50 (0.136)
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Treatment comparison: Vadadustat minus Darbepoetin Alfa; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Least squares mean difference = -0.07, 95% CI 2-sided [-0.34 to 0.19], Standard Error of Mean 0.134

4. Secondary Outcome: Median Time to First MACE Plus Hospitalization for Heart Failure or Thromboembolic Event Excluding Vascular Access Thrombosis
Description: MACE was defined as all-cause mortality, non-fatal MI, or non-fatal stroke. Hospitalization for EAC adjudicated heart failure included presentation of participants to an acute care facility requiring an overnight hospitalization (change in calendar day) with an exacerbation of heart failure requiring treatment. EAC confirmed thromboembolic events for this secondary outcome measure included arterial thrombosis, deep vein thrombosis, and pulmonary embolism. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0016 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 176 weeks
Population: Safety Population (INNO2VATE). Only those participants with MACE plus hospitalization for heart failure or thromboembolic event excluding vascular access thrombosis were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 29 | 31
Weeks | 27.14 [14.14 to 46.14] | 47.00 [21.86 to 61.57]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0016 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.8871, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.618 to 1.743]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first MACE plus hospitalization for heart failure or thromboembolic event Excluding vascular access thrombosis for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 420 and 449 respectively; median time to first event (Q1, Q3) = 42.07 (21.50, 71.14) weeks versus 45.29 (22.29, 72.43) weeks, respectively; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.4096, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.840 to 1.096]

5. Secondary Outcome: Median Time to First Cardiovascular MACE
Description: MACE was defined as all-cause mortality, non-fatal MI, or non-fatal stroke. Cardiovascular MACE analysis differed from the primary MACE endpoint as it included only deaths adjudicated by the EAC as cardiovascular deaths (i.e, only EAC-confirmed cardiovascular deaths) in addition to first events of non-fatal MI or non-fatal stroke. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0016 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 176 weeks
Population: Safety Population (INNO2VATE). Only those participants with cardiovascular MACE events were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 16 | 14
Weeks | 18.50 [11.29 to 34.43] | 54.07 [35.29 to 67.00]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0016 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.5210, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.670 to 2.771]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first cardiovascular MACE for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 225 and 242 respectively; median time to first event (Q1, Q3) = 43.29 (21.71, 77.14) weeks versus 45.79 (21.14, 73.86) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.5007, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.795 to 1.144]

6. Secondary Outcome: Median Time to First Cardiovascular Death
Description: Cardiovascular death included EAC adjudicated fatal MI, pump failure, sudden death, presumed sudden death, fatal stroke, fatal pulmonary embolism, cardiovascular procedure-related death, other cardiovascular death, and presumed cardiovascular death. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0016 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 176 weeks
Population: Safety Population (INNO2VATE). Only those participants with cardiovascular death were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 9 | 10
Weeks | 22.00 [12.71 to 33.14] | 58.14 [21.86 to 67.57]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0016 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.9527, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.452 to 2.666]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first cardiovascular death for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 150 and 160 respectively; median time to first event (Q1, Q3) = 43.71 (27.43, 77.14) weeks versus 49.29 (24.43, 74.07) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.6284, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.766 to 1.195]

7. Secondary Outcome: Median Time to First All-cause Mortality
Description: Only events that were positively adjudicated and confirmed by the EAC were included in the MACE analyses. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0016 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 176 weeks
Population: Safety Population (INNO2VATE). Only those participants with all-cause mortality were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 15 | 20
Weeks | 31.71 [13.71 to 62.00] | 45.36 [21.57 to 58.14]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0016 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.5115, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.388 to 1.555]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first all-cause mortality for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 291 and 310 respectively; median time to first event (Q1, Q3) = 50.00 (29.71, 79.00) weeks versus 49.57 (25.86, 77.29) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.4878, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.812 to 1.118]

8. Other Pre Specified Outcome: Exploratory - Proportion of Participants With Hb Values Within the Target Range During the Primary Evaluation Period (Weeks 24 to 36)
Time Frame: Weeks 24 to 36
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory - Proportion of Time With Hb Values Within the Target Range During the Primary Evaluation Period (Weeks 24 to 36)
Time Frame: Weeks 24 to 36
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory - Proportion of Time With Hb Values Within the Target Range During the Secondary Evaluation Period (Weeks 40 to 52)
Time Frame: Weeks 40 to 52
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory - Proportion of Participants With Hb Values Within the Target Range During the Secondary Evaluation Period (Weeks 40 to 52)
Time Frame: Weeks 40 to 52
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory - Proportion of Participants With an Hb Increase of >1.0 g/dL From Baseline Visit
Time Frame: Baseline; up to Week 52
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory - Time to Achieve Hb Increase of >1.0 g/dL From Baseline Visit
Time Frame: Baseline; up to Week 52
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Exploratory - Mean Change in Hb Between Baseline (Mean Pretreatment Hb) and the Primary Evaluation Period (Mean Hb From Weeks 24 to 36) Stratified by Pre-baseline Erythropoiesis-stimulating Agent (ESA) Exposure
Time Frame: Baseline; Weeks 24 to 36
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Exploratory - Mean Monthly Dose of Intravenous (IV) Elemental Iron Administered in Participants Who Have Received IV Iron
Time Frame: Up to Week 52
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exploratory - Proportion of Participants Receiving IV Iron Therapy
Time Frame: Up to Week 52
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Exploratory - Proportion of Participants Receiving Red Blood Cells (RBCs) Transfusion(s)
Time Frame: Up to Week 52
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 176 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported in study AKB-6548-CI-0016 (NCT02865850). Of the participants randomized, 365 participants were included in the Safety population (179 and 186 participants in the Vadadustat and Darbepoetin alfa treatment groups, respectively). Four randomized participants did not receive treatment.
Arm/Group | Vadadustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 15/179 | 20/186
Serious Adverse Events (participants affected / at risk) | 89/179 | 105/186
Other Adverse Events (participants affected / at risk) | 79/179 | 83/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=179) | Darbepoetin Alfa (N=186)
Pneumonia (Infections and infestations) | 8 | 7
Fluid overload (Metabolism and nutrition disorders) | 10 | 2
Hypertensive urgency (Vascular disorders) | 7 | 3
Sepsis (Infections and infestations) | 3 | 6
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Coronary artery disease (Cardiac disorders) | 4 | 4
Osteomyelitis (Infections and infestations) | 4 | 4
Acute myocardial infarction (Cardiac disorders) | 3 | 4
Atrial fibrillation (Cardiac disorders) | 3 | 4
Cardiac failure congestive (Cardiac disorders) | 3 | 4
Non-cardiac chest pain (General disorders) | 3 | 3
Cellulitis (Infections and infestations) | 4 | 2
Gangrene (Infections and infestations) | 3 | 3
Peritonitis (Infections and infestations) | 3 | 3
Staphylococcal sepsis (Infections and infestations) | 4 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cardiac arrest (Cardiac disorders) | 2 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypertension (Vascular disorders) | 2 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 2 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 4
Device related infection (Infections and infestations) | 3 | 1
Hepatitis B (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 1 | 3
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 | 3
Alanine aminotransferase increased (Investigations) | 1 | 3
Pulseless electrical activity (Cardiac disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Arteriovenous fistula site infection (Infections and infestations) | 1 | 2
Device related sepsis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 2
Vascular device infection (Infections and infestations) | 1 | 2
Hepatic enzyme increased (Investigations) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 2
Cardiogenic shock (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 2 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Complication associated with device (General disorders) | 0 | 2
Death (General disorders) | 1 | 1
Impaired healing (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Acute hepatitis B (Infections and infestations) | 1 | 1
Arteriovenous graft site infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Renal graft infection (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Transaminases increased (Investigations) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 1 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Arteriosclerosis (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Blood disorder (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Angle closure glaucoma (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Retinal artery thrombosis (Eye disorders) | 0 | 1
Abdominal migraine (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Dolichocolon acquired (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Cardiac death (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 0 | 1
Porcelain gallbladder (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 0 | 1
Catheter site abscess (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Cytomegalovirus syndrome (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Osteomyelitis acute (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Renal cyst infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Serratia bacteraemia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Subacute endocarditis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Vascular access site infection (Infections and infestations) | 1 | 0
Wound abscess (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Brain stem syndrome (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebral hypoperfusion (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Postresuscitation encephalopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Brachiocephalic vein thrombosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
Steal syndrome (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=179) | Darbepoetin Alfa (N=186)
Hypertension (Vascular disorders) | 27 | 24
Diarrhoea (Gastrointestinal disorders) | 18 | 17
Nausea (Gastrointestinal disorders) | 14 | 13
Urinary tract infection (Infections and infestations) | 9 | 16
Procedural hypotension (Injury, poisoning and procedural complications) | 11 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Vomiting (Gastrointestinal disorders) | 13 | 9
Hypotension (Vascular disorders) | 5 | 16
Dialysis related complication (Injury, poisoning and procedural complications) | 8 | 11
Headache (Nervous system disorders) | 8 | 11
Nasopharyngitis (Infections and infestations) | 10 | 8
Fall (Injury, poisoning and procedural complications) | 10 | 8
Constipation (Gastrointestinal disorders) | 3 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT02865850/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT02865850/SAP_001.pdf